CLINICAL TRIAL: NCT01066481
Title: A Phase 2, Multi-Center, Double-Blinded, Placebo-Controlled Safety And Efficacy Study Of Oral PF-01913539 In Patients With Mild To Moderate Alzheimer's Disease
Brief Title: A Study Of Oral PF-01913539 In Patients With Mild To Moderate Alzheimer's Disease
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B1451010
Record Dates: First submitted 2010-02-09; First posted 2010-02-10 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2010-06

CONDITIONS: Alzheimer's Disease; Dementia; Dimebon; Investigational Drug
Keywords: Alzheimer's disease; clinical trial; memory loss; investigational drug; neurodegenerative disease; dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia; Memory Disorders; Neurodegenerative Diseases | interventions — latrepirdine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PF-01913539 5 mg three times daily (Experimental): PF-01913539 5 mg three times daily for 6 months
  Interventions: Drug: PF-01913539 5 mg
- PF-01913539 20 mg three times daily (Experimental): PF-01913539 20 mg three times daily for 6 months
  Interventions: Drug: PF-01913539 5 mg
- Placebo (Placebo Comparator): Placebo three times daily for 6 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-01913539 5 mg — PF-01913539 5 mg three times daily for 6 months
  Arms: PF-01913539 5 mg three times daily
Drug: PF-01913539 5 mg — PF-01913539 5 mg three times daily for 6 months
  Arms: PF-01913539 20 mg three times daily
Drug: Placebo — Placebo three times daily for 6 months
  Arms: Placebo

SUMMARY:
The purpose of this study is to demonstrate the safety and efficacy of PF-01913539 in the treatment of patients with mild-to-moderate Alzheimer's Disease. It is a 6-month study enrolling 651 patients in Japan, Hong Kong, Korea, and Republic of China. All patients completing the 6-month study will be eligible to receive PF-01913539 in an open-label extension trial (B1451031).

ELIGIBILITY:
Inclusion Criteria:

* Mild-to-Moderate Alzheimer's disease
* MMSE score 10-24 inclusive

Exclusion Criteria:

* Administration of anti-dementia drugs including cholinesterase-inhibitors or NMDA receptor antagonists within 90 days
* Complication of other causes of dementia

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-04; Primary Completion 2012-03 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Mean change in the Alzheimer's Disease Assessment Scale Cognitive Subscale (ADAS-cog) score from baseline. | 26 weeks
Distribution of Clinician's Interview-Based Impression of Change plus Caregiver (CIBIC-plus) Input | 26 weeks

SECONDARY OUTCOMES:
Mean change in Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADAS-ADL) score from baseline. | 12, 26 weeks
Mean change in Neuropsychiatric Inventory (NPI) score from baseline. | 12, 26 weeks
Mean change in Mini-Mental State Examination (MMSE) score from baseline. | 6, 12, 18, 26 weeks
Mean change in each item of Resource Utilization In Dementia(RUD) Lite from baseline. | 12, 26 weeks
Adverse events, physical examination, vital signs (blood pressure, temperature, and heart rate), 12-lead ECG, and laboratory tests (hematology, blood chemistry and urinalysis). | 12, 26 weeks
Population PK parameters (CL/F, V/F, etc.) | 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1451010&StudyName=A%20Study%20Of%20Oral%20PF-01913539%20In%20Patients%20With%20Mild%20To%20Moderate%20Alzheimer%27s%20%20Disease